CLINICAL TRIAL: NCT05937542
Title: A Qualitative Investigation of the Experiences of Participants Undertaking a CycLing and EducATional (CLEAT) Programme for the Treatment of Hip Osteoarthritis.
Brief Title: A Qualitative Investigation of CLEAT Participants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bournemouth University (Other)
Collaborators: Economic and Social Research Council, United Kingdom (Other)
Responsible Party: Sponsor
Other Study IDs: 330860
Record Dates: First submitted 2023-06-27; First posted 2023-07-10 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Qualitative Investigation of Participant Experiences — There is no intervention. This is a retrospective qualitative study.

SUMMARY:
As the United Kingdom's National Health Service (NHS) waiting list soars above seven million people, with treatment wait times over two years, older people with chronic conditions face worsening symptoms, increased use of medications, more complicated surgeries with slower recovery, reduced quality of life, and loss of independence. As part of its plans to tackle this crisis, the NHS promotes exercise as a "miracle cure" for arresting the progress of disease and helping disease management and recovery. However, current plans promoting individual, home-based exercise, as well as on-site hospital-based programs of delivery, have met with only limited success, and face problems of decreased space, capacity, clinician time, as well as lack of knowledge and expertise with regard to effective behavior change. We have developed a community-based group exercise programme for older people with hip osteoarthritis. This community-based group exercise programme has successfully helped those with hip osteoarthritis (3.5 million over 45s in the UK) reduce pain and need for medication, as well as avoiding surgery, and has formed part of an NIHR trial examining the use of exercise and education versus standard physiotherapy care for the treatment of hip osteoarthritis. In order to better understand the mechanisms of action of this programme, the present study will examine, via focus groups interviews, the experiences of participants who have undertaken the exercise and education programme. The data generated from the focus groups will help to elucidate what "works" within the programme and will help inform future development of resources to support health professionals in providing exercise rehabilitation for older people with chronic conditions.

ELIGIBILITY:
Inclusion Criteria:

Participants who had previously been part of the NIHR-funded CLEAT trial. Those participants were defined as follows:

* Diagnosed with osteoarthritis of the hip as per NICE criteria.
* Male and female, aged 45 years and over
* Meeting the GP criteria for exercise referral
* Capable of giving informed consent
* Be able to understand English as necessary to benefit from the intervention, in the investigators' opinion.

Exclusion Criteria:

• Anyone not previously part of the NIHR-funded CLEAT trial. -

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who had previously been part of the NIHR-funded trial into the effects of a cycling and educational intervention for people with hip osteoarthritis.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Participant Experiences | One data collection point via interview (3-6 months)
  Participant experiences generated via qualitative data

CONTACTS AND LOCATIONS:
Overall Officials: Tim Rees, PhD, Study Director — Professor in Sport
Locations (1):
- Bournemouth University, Bournemouth, United Kingdom